CLINICAL TRIAL: NCT03150069
Title: Pregnancy With Morquio Syndrome - What Are Patients' Perspectives and Has ERT Changed Them?
Acronym: MorqPreg
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Nadia Ali, PhD, Principal Investigator, Emory University
Other Study IDs: IRB00088777
Record Dates: First submitted 2017-05-10; First posted 2017-05-11 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Morquio Disease; MPS - Mucopolysaccharidosis
Keywords: Pregnancy
MeSH Terms: conditions — Mucopolysaccharidosis IV; Mucopolysaccharidoses | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Morquio A / Biological Mothers: Women with Morquio A who have biological children
  Interventions: Other: Interview
- Morquio A / No Biological Children: Women with Morquio A who do not have biological children (both adoptive mothers and non-mothers)
  Interventions: Other: Interview
- Morquio B / Biological Mothers: Women with Morquio B who have biological children
  Interventions: Other: Interview
- Morquio B / No Biological Children: Women with Morquio B who do not have biological children (both adoptive mothers and non-mothers)
  Interventions: Other: Interview

INTERVENTIONS:
Other: Interview — In-person or telephone in-depth interview

SUMMARY:
The present study seeks to interview women with Morquio A and Morquio B syndrome, to explore their concerns surrounding pregnancy and the impact of ERT on their perspectives, in comparison with the control group of Morquio B subjects for whom no ERT treatment exists.

Interviews will be conducted by a health psychologist, in-person or over the telephone. Data will be analyzed using MAXQDA 12.0 software and Grounded Theory. Differences in thematic trends between Morquio A subjects, for whom treatment exists, and a control group of Morquio B subjects, for whom there is no treatment, will be compared.

DETAILED DESCRIPTION:
The present study seeks to interview women with Morquio A and Morquio B syndrome themselves, to explore and discover their perspectives and concerns surrounding pregnancy and having biological children, the impact of the advent of ERT for Morquio A on their perspectives and concerns in comparison with the control group of Morquio B subjects for whom no ERT treatment exists, as well as what each group is being told by the medical community and others in their lives in this regard.

Interviews will be conducted by a health psychologist, either in-person or over the telephone. We will interview 1) those women with Morquio syndrome who are known to have been pregnant and 2) those women with Morquio syndrome who have not been pregnant and/or chose to adopt children. All information will be kept confidential, except as in accordance with Georgia law relating to reporting of child or elder abuse, suicidal and/or homicidal intent.

Data will be analyzed using MAXQDA 12.0 software to develop code which can be used to describe and compare the data using Grounded Theory. Differences in thematic trends between Morquio A subjects, for whom treatment exists, and a control group of Morquio B subjects, for whom there is no treatment, will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Documented clinical diagnosis of either MPS IVA or MPS IVB, based on clinical signs and symptoms, documented reduced fibroblast or leukocyte GALNS enzyme activity or genetic testing confirming diagnosis.
2. Subject is at least 15 years old.
3. Subject is female.
4. Subject is fluent enough in English to complete in-depth interview with PI.

Exclusion Criteria:

1. Patient has a clinically significant disease other than Morquio which would confound the effects of Morquio upon study variables.
2. Any condition that, in the view of the Investigator, places the patient at high risk of poor compliance or of not completing the study.

Ages: 15 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Women with Morquio syndrome, at least 15 years of age, English-speaking
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2018-08-17 (Actual)

PRIMARY OUTCOMES:
Completion of in-depth interview | Approximately 1 hour
  Completion of in-depth interview

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Decatur, Georgia, United States

IPD SHARING:
Plan to Share IPD: No